CLINICAL TRIAL: NCT01504529
Title: Non-Interventional, Retrospective, Multi-center Study to Evaluate Non-Motor Symptoms in Advanced PD Patients Already Treated With Rotigotine
Brief Title: Non-interventional, Retrospective, Multi-center Study to Evaluate Non-motor Symptoms in Advanced Parkinson Disease (PD) Patients Already Treated With Rotigotine
Acronym: RETO-PD
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Collaborators: Pivotal S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: SP1018; UCB-ROT-2011-01
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Parkinson's Disease
Keywords: Rotigotine (Neupro); Non-Motor Symptoms; Advanced Parkinson's Disease; Local study; Spain; Observational study; Non-interventional study; Retrospective study; Post-marketing study; Multicenter study
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neupro Treatment: Data from patients with advanced PD who have been treated with Rotigotine (Neupro®) for at least the previous 6 months as prescribed by physicians according to usual clinical practice in Spain, will be retrospectively collected.

SUMMARY:
This is an observational, non-interventional and retrospective study in patients with advanced PD who have been treated with Rotigotine (Neupro®) as prescribed by physicians according to usual clinical practice in Spain.

The Primary Objective will be to evaluate Non-Motor Symptoms (NMS) in advanced PD patients who have been treated with Rotigotine for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, all of the following criteria must be met:

* Male and female ambulatory patients with Parkinson's disease diagnosis (as per the London Brain Bank diagnosis criteria) ≥6 months ago
* Patient aged 30 years or older at the time of Parkinson's disease diagnosis
* Patients who were under treatment with Rotigotine following routine clinical practice, either alone or in combination with Levodopa, and in an advanced PD dosage (≥ 8 mg/ 24 h) for at least the previous 6 months
* Patients under treatment with Rotigotine (≥ 8 mg/ 24 h) who were assessed twice of NMS by means of the PDNMS-Q 6 months apart
* Patients are currently informed and have been given enough time and opportunity to think about participation (data collection) in the study and have given written informed consent

Exclusion Criteria:

Patients are not permitted to enroll in the study if any of the following criteria is met during the previous 6 months:

* Patients have other Parkinsonian syndrome different than Parkinson´s disease
* Patients have a history of Pallidotomy, Thalamotomy, Deep Brain Stimulation or Fetal Tissue Transplant
* Patients with Dementia, active Hallucinations or active or treated Psychosis
* Patients with any other neurological / psychological disorder
* Patients who had received Central Nervous System (CNS) active therapy (e.g. sedatives, hypnotics, anti-depressants, anxiolytics, atypical neuroleptics, etc)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As a retrospective Observational Study, the data will be obtained from the medical records of the patients with advanced PD who have been treated for at least 6 months with Rotigotine (Neupro®) as prescribed by physicians according to usual clinical practice in Spain.
  The study will approximately include 400 patients from 80 Spanish sites.
Sampling Method: Non-Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Month 6 in Non-Motor Symptoms (NMS) as assessed by the Parkinson's Disease Non-Motor Symptoms Questionnaire (PDNMS-Q) | From Baseline to Month 6

SECONDARY OUTCOMES:
Change from Baseline to Month 6 in Unified Parkinson's Disease Rating Scale (UPDRS) Part III | From Baseline to Month 6
Change from Baseline to Month 6 in Hoehn & Yahr stage | From Baseline to Month 6

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (59):
- Spain (59):
  - 65, A Coruña
  - 66, A Coruña
  - 68, A Coruña
  - 33, Albacete
  - 25, Alicante
  - 26, Alicante
  - 27, Alicante
  - 14, Avilés
  - 17, Baleares
  - 42, Barcelona
  - 43, Barcelona
  - 44, Barcelona
  - 45, Barcelona
  - 47, Barcelona
  - 48, Barcelona
  - 49, Barcelona
  - 52, Barcelona
  - 85, Barcelona
  - 58, Bera
  - 55, Bilbao
  - 10, Cadiz
  - 32, Ciudad Real
  - 34, Cuenca
  - 53, Girona
  - 59, Guipúzcoa
  - 11, Huesca
  - 16, Islas Baleares
  - 3, Jaén
  - 4, Jaén
  - 50, Lleida
  - 69, Lugo
  - 70, Madrid
  - 71, Madrid
  - 73, Madrid
  - 74, Madrid
  - 75, Madrid
  - 76, Madrid
  - 78, Madrid
  - 79, Madrid
  - 80, Madrid
  - 18, Maó
  - 15, Mieres
  - 81, Murcia
  - 82, Murcia
  - 83, Navarra
  - 13, Oviedo
  - 63, Pontevedra
  - 67, Pontevedra
  - 29, Santa Cruz de Tenerife
  - 30, Santa Cruz de Tenerife
  - 31, Santa Cruz de Tenerife
  - 38, Segovia
  - 36, Toledo
  - 19, Valencia
  - 20, Valencia
  - 22, Valencia
  - 23, Valencia
  - 24, Valencia
  - 56, Vizcaya

REFERENCES:
- [Derived] Valldeoriola F, Salvador A, Gomez-Arguelles JM, Marey J, Moya M, Ayuga A, Ramirez F. The effects of transdermal rotigotine on non-motor symptoms of Parkinson's disease: a multicentre, observational, retrospective, post-marketing study. Int J Neurosci. 2018 Apr;128(4):369-375. doi: 10.1080/00207454.2017.1387111. Epub 2017 Dec 17. PMID 29249180